CLINICAL TRIAL: NCT03245034
Title: Assessing the Impact of Acupuncture Therapy on Medical Resident Well-Being: Feasibility and Acceptance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-02292
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Exhaustion; Syndrome
Keywords: Medical Residents; Well-Being; Stress/Burnout in Medical Residents
MeSH Terms: conditions — Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fourth-year Obstetrics and Gynecology residents (Experimental): The intervention will be three sessions of auricular acupuncture therapy; there will be no control intervention.
  Interventions: Behavioral: Auricular Acupuncture Therapy

INTERVENTIONS:
Behavioral: Auricular Acupuncture Therapy — Acupuncture treatment will be the NADA protocol, a well-known and commonly used protocol that has previously been studied for stress relief in health care workers.In this protocol, 5, ½" needles are inserted in each auricle and retained while the group relaxes for 20 minutes. It will be conducted by two acupuncturists credentialed at NYU Lutheran (TK and AG).

SUMMARY:
This feasibility study develops methods for larger-scale research, evaluating the acceptability and perceived impact of a group acupuncture and acupressure intervention, as well as suitability of a self-report instrument. During their weekly training program, eleven OB residents at NYU Lutheran Medical Center will receive three sessions of auricular acupuncture therapy. (This resident population was previously anonymously surveyed and all expressed interest in participating in such a study). The Professional Quality of Life Scale (ProQOL) will be administered at 6 time points. A brief survey will also be given to assess participants' acceptance of the intervention as well as applicability of the ProQOL instrument. Additional feasibility-related outcomes include protocol compliance/withdrawals, adverse events, and time taken to complete intervention and surveys.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in NYU Lutheran Obstetrics & Gynecology Residency program

Exclusion Criteria:

* Women currently pregnant or attempting to conceive

Ages: 25 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Professional Quality of Life (ProQOL) | 4 Weeks
  he ProQOL is the most commonly used measure of the negative and positive affects of helping others who experience suffering and trauma. The ProQOL has sub-scales for compassion satisfaction, burnout and compassion fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Meera Kesavan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided